CLINICAL TRIAL: NCT00373932
Title: Real-Time Support for Exercise Persistence in COPD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Huong Q. Nguyen, PhD, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 29494-V2; R03NR009361-01A1 (NIH)
Record Dates: First submitted 2006-09-06; First posted 2006-09-08 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive; COPD; Emphysema; Chronic Bronchitis
Keywords: Exercise; Physical Activity; Adherence
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MOBILE-A (Experimental): Coached exercise persistence intervention
  Interventions: Behavioral: Coached exercise persistence intervention
- MOBILE-B (Active Comparator): Self-monitored exercise persistence intervention
  Interventions: Behavioral: Self-Monitored exercise persistence intervention

INTERVENTIONS:
Behavioral: Coached exercise persistence intervention — Collaborative symptom and exercise monitoring and weekly reinforcement for exercise persistence from nurse coach via a mobile device and telephone.
  Arms: MOBILE-A
Behavioral: Self-Monitored exercise persistence intervention — Self-monitoring of symptoms and exercise using a mobile device
  Arms: MOBILE-B

SUMMARY:
The purpose of this exploratory study is to determine the feasibility, acceptability, and efficacy of an exercise persistence intervention for patients with chronic obstructive pulmonary disease (COPD) following pulmonary rehabilitation (PR).

DETAILED DESCRIPTION:
Exercise, a cornerstone of PR, is effective in improving dyspnea, functioning, and health related quality of life (HRQL) in patients with COPD. However, these improvements gradually dissipate following program completion. There are currently few successful interventions that support patients' persistence with community-based exercise after PR and that have closely monitored the potentially negative impact that COPD exacerbations have on exercise behaviors. Emerging technologies such as wirelessly enabled personal digital assistants (PDA) may provide an innovative means to support exercise persistence through real-time collaborative monitoring of exercise and signs and symptoms of COPD exacerbations and reinforcement to enhance exercise self-efficacy. Patient graduates of two PR programs who have COPD (n=20) will first undergo a 2-week run-in prior to being randomized to either the MOBILE (Mobilizing Support for Long-term Exercise) intervention or attention control for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe COPD (FEV1/FVC <70% and FEV1%<80%)
* Ability to speak, read and write English
* Age 40 or older
* Willingness to complete a 6 month program

Exclusion Criteria:

* Illnesses such as bronchiectasis, active malignancies or other end stage diseases
* Plans to continue in a maintenance program after rehabilitation.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Exercise behavior | 3 & 6 Months

SECONDARY OUTCOMES:
Self-efficacy for exercise | 3 & 6 Months
Perception of support | 3 & 6 Months
COPD exacerbation | 3 & 6 Months
Exercise Performance | 3 & 6 months
Health related quality of life | 3 & 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Huong Q. Nguyen, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Nguyen HQ, Steele BG, Dougherty CM, Burr RL. Physical activity patterns of patients with cardiopulmonary illnesses. Arch Phys Med Rehabil. 2012 Dec;93(12):2360-6. doi: 10.1016/j.apmr.2012.06.022. Epub 2012 Jul 5. PMID 22772084
- [Derived] Nguyen HQ, Gill DP, Wolpin S, Steele BG, Benditt JO. Pilot study of a cell phone-based exercise persistence intervention post-rehabilitation for COPD. Int J Chron Obstruct Pulmon Dis. 2009;4:301-13. doi: 10.2147/copd.s6643. Epub 2009 Sep 1. PMID 19750190